CLINICAL TRIAL: NCT00807963
Title: Phase I, Open-Label, Pharmacokinetic, Safety and Tolerability Study of Subcutaneously Administered Bisphosphonate With Recombinant Human Hyaluronidase (rHuPH20) vs Bisphosphonate
Brief Title: Pharmacokinetic, Safety and Tolerability Study of SC Administered Bisphosphonate With rHuPH20 vs Bisphosphonate Alone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Halozyme Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: HZ2-08-02
Record Dates: First submitted 2008-12-11; First posted 2008-12-15 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Risk Factors for or a Diagnosis of Osteoporosis
Keywords: Pharmacokinetics; rHuPH20
MeSH Terms: interventions — Zoledronic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- Stage 1: rHuPH20 plus ZA (Experimental): Participants will receive one of several dose/concentrations of recombinant human hyaluronidase PH20 (rHuPH20) with zoledronic acid (ZA).
  Interventions: Drug: rHuPH20; Drug: zoledronic acid
- Stage 2: ZA (Experimental): Participants will receive a dose/concentration of ZA administered without rHuPH20.
  Interventions: Drug: zoledronic acid
- Stage 3: rHuPH20 plus ZA (Experimental): Participants will receive one of several dose/concentrations of rHuPH20 with ZA.
  Interventions: Drug: rHuPH20; Drug: zoledronic acid
- Stage 4: ZA (Experimental): Participants will receive an intravenous (IV) dose of 5 milligrams (mg) ZA.
  Interventions: Drug: zoledronic acid
- Stage 4: ZA with rHuPH20 (Experimental): Participants will receive a subcutaneous (SC) dose of ZA with rHuPH20.
  Interventions: Drug: rHuPH20; Drug: zoledronic acid

INTERVENTIONS:
Drug: rHuPH20 — recombinant human hyaluronidase PH20 injection
  Arms: Stage 1: rHuPH20 plus ZA; Stage 3: rHuPH20 plus ZA; Stage 4: ZA with rHuPH20
Drug: zoledronic acid — subcutaneous injection

SUMMARY:
The purpose of this study is to determine the maximum tolerated concentration (MTC) of bisphosphonate with a fixed dose of rHuPH20 administered SC, the MTC of bisphosphonate without rHuPH20 administered SC, the optimal dose of rHuPH20 to deliver bisphosphonate SC at MTC, and to compare the PK of SC administered bisphosphonate at MTC with optimal dose rHuPH20 to bisphosphonate alone.

ELIGIBILITY:
Inclusion Criteria:

* Male or female volunteers 18 to 60 years of age, inclusive.
* Intact normal skin in the area intended for administration.
* Adequate venous access in both upper extremities.
* Dental examination by an appropriately trained professional within 14 days of administration demonstrating no signs, symptoms, or risk factors of osteonecrosis of the jaw (ONJ).
* Vital signs (BP, HR, temperature, respiratory rate) within normal range or, if out of range, assessed by the Investigator as not clinically significant and it is mutually agreed by both Investigator and Sponsor Medical Monitor that the subject need not be excluded from the study for this reason.
* Electrocardiogram within normal range or if out of range, assessed by the Investigator as not clinically significant and it is mutually agreed by both Investigator and Sponsor Medical Monitor that the subject need not be excluded from the study for this reason.
* Within 14 days prior to administration, metabolic panel (e.g., sodium, potassium, chloride, bicarbonate, BUN, creatinine, glucose, calcium, AST, ALT, alkaline phosphatase, total bilirubin, albumin, and total protein) and complete blood count within the laboratory normal reference range or, if out of range, assessed by the Investigator as not clinically significant and it is mutually agreed by both Investigator and Sponsor Medical Monitor that the subject need not be excluded from the study for this laboratory value.
* A negative serum or urine pregnancy test (if female of child-bearing potential) within 14 days of study drug administration.
* Female subjects of child-bearing potential must agree to be currently practicing effective birth control or abstinence and agree to continue to do so for at least 30 days after duration of their time on study.
* Decision-making capacity and willingness and ability to comply with the requirements for full completion of the trial.
* Signed, written IRB/EC-approved informed consent.

Exclusion Criteria:

* Lower extremity edema.
* Lower extremity pathology that could interfere with any protocol-specified outcome assessment (e.g., cellulitis, lymphatic disorder or prior surgery, pre-existing pain syndrome, auxiliary lymph node dissection, etc.).
* Creatinine clearance < 60 mL/min (Cockcroft-Gault formula).
* Any risk factor for bisphosphonate-related renal toxicity including by not limited to known predisposition to or history of renal insufficiency or renal failure, hypertension, diabetes mellitus, volume depletion, sepsis, paraproteinemia, and subjects receiving known nephrotoxic drugs.
* Dehydration Grade 2 or higher based on NCI CTCAE V3.0.
* Known parathyroid gland dysfunction or any other disease that could lower blood calcium levels.
* Known history and/or electrocardiographic evidence of atrial fibrillation.
* Known allergy to any hyaluronidase.
* Bisphosphonate treatment within preceding six months.
* Known allergy or intolerance to any bisphosphonate.
* Pregnancy or breast-feeding woman.
* Known clinically significant cardiovascular, gastrointestinal, hepatic, neurological, psychiatric, endocrine, cancer, HIV infection, diabetes mellitus, intercurrent illness such as influenza, or other major systemic disease that would unduly risk the subject's safety or interfere with the interpretation of results.
* Participation in a study of any investigational drug or device within 30 days of enrollment in this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2008-12; Primary Completion 2009-09-21 (Actual); Study Completion 2009-09-21 (Actual)

PRIMARY OUTCOMES:
Assessment of local tolerability of injected drug product | Over a 7 day period

CONTACTS AND LOCATIONS:
Overall Officials: Emanuel P DeNoia, MD, Principal Investigator — Healthcare Discoveries, LLC/ICON
Locations (1):
- Healthcare Discoveries, LLC/ICON Development Solutions, San Antonio, Texas, United States